CLINICAL TRIAL: NCT00072501
Title: Screening Breast Ultrasound in High-Risk Women
Brief Title: Breast Ultrasound and Mammography in Screening Women at High Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Screening
Other Study IDs: CDR0000339812; ACRIN-6666
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2006-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

INTERVENTIONS:
Procedure: breast imaging study
Procedure: comparison of screening methods
Procedure: magnetic resonance imaging
Procedure: radiomammography
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Screening tests such as ultrasound and mammography may help doctors detect cancer cells early and plan more effective treatment for breast cancer. It is not yet known whether ultrasound is more effective than mammography in detecting breast cancer.

PURPOSE: This clinical trial is studying breast ultrasound to see how well it works compared to mammography in detecting cancer in women who are at high risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the diagnostic yield of whole breast bilateral screening ultrasound and mammography for the detection of breast cancer in women at high risk for breast cancer.
* Determine the cancer detection yield of a single contrast-enhanced magnetic resonance imaging (MRI) examination after 3 rounds of annual screening with ultrasound and mammography in these participants. (MRI component of the study)

Secondary

* Determine the independent sensitivity and specificity of these screening methods in these participants.
* Correlate performance of these screening methods with selected participant characteristics (e.g., breast density and heterogeneity of the parenchyma).
* Validate the sonographic classification of lesions as "probably benign" and estimate the rate of malignancy in participants screened with these methods.
* Determine the cost effectiveness associated with screening breast ultrasound, in terms of radiologist and resource time performing the exam and the induced cost of screening ultrasound (e.g., follow-up and biopsy).
* Determine the reproducibility of lesion identification, measurement of lesion diameters, and volume and recording of lesion location on ultrasound in these participants.
* Determine the size, type, grade, and nodal status of cancers seen only on MRI in these participants. (MRI component of the study)
* Estimate the rate of benign biopsies and short interval follow-up induced only by MRI in these participants. (MRI component of the study)
* Determine the cost effectiveness of MRI, including induced costs of unnecessary biopsies and follow-up. (MRI component of the study)
* Compare the agreement among multiple examiners in sonographic, mammographic, and MRI feature analysis (using terms from the BI-RADS® lexicon) and final assessment (e.g., estimated probability of malignancy and/or recommendation for biopsy) in the enriched set of diagnostic training cases with consensus and histopathologic reference standards.

OUTLINE: This is a randomized, multicenter study. Participants are randomized to 1 of 2 screening arms.

* Arm I: Participants undergo physician-performed bilateral whole breast ultrasound (US) followed by mammogram within 2 weeks.
* Arm II: Participants undergo mammogram followed by physician-performed bilateral whole breast US within 2 weeks.

In both arms, participants with negative or benign findings are rescreened according to their screening arm at 1 and 2 years. Participants with "probably benign" findings are rescreened at the 6-month follow-up visit. Participants with findings that are suspicious or highly suggestive of malignancy are recommended for biopsy.

A subset of participants* in both arms undergo contrast-enhanced breast MRI within 4 weeks after completion of the 2-year screening US and mammogram. Participants with "probably benign" findings seen only on MRI may undergo an additional breast MRI at the 6-month follow-up visit. Participants with additional suspicious lesions seen only on MRI undergo second-look targeted US for biopsy guidance or MRI-guided vacuum-assisted biopsy after completion of any biopsies or additional views prompted by the 2-year screening US and mammogram visit.

NOTE: *No diagnosis of metastatic cancer of any type since entering this clinical trial.

Participants are followed annually for 3 years.

PROJECTED ACCRUAL: A total of 2,808 participants will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At high risk for breast cancer, as defined by at least 1 of the following:

  * Known BRCA1 or BRCA2 mutation
  * Personal history of breast cancer with conserved breast analyzed separately
  * Prior biopsy showing atypical ductal hyperplasia, atypical lobular hyperplasia, or atypical papilloma and not receiving chemoprevention (i.e., not on tamoxifen, raloxifene, anastrazole, or any other aromatase inhibitor) OR any of these atypical lesions (including phyllodes tumors) AND first-degree relative diagnosed with breast cancer under age 50
  * Prior biopsy showing lobular carcinoma in situ
  * Age 30 and under and received prior chest and/or mediastinal and/or axillary irradiation ≥ 8 years ago
  * Risk of breast cancer meeting one of the following criteria:

    * Gail or Claus lifetime cancer risk ≥ 25%
    * Gail 5-year cancer risk ≥ 2.5%
    * Gail 5-year cancer risk ≥ 1.7% AND known to have extremely dense breasts (≥ 75% dense) by most recent mammogram
* Heterogeneously dense (≥ 50% dense) or extremely dense (≥ 75% dense throughout the entire breast) breast parenchyma in at least 1 breast by mammogram* OR unknown breast density due to no prior mammogram NOTE: *No fatty breasts or minimal scattered fibroglandular density
* Most recent mammogram* (if any) was interpreted as negative, benign, and/or remarkable only for post-treatment changes NOTE: *At least 11 full months since prior mammogram
* No current signs or symptoms of breast cancer (e.g., palpable breast masses, bloody or spontaneous clear nipple discharge, axillary mass, or abnormal skin changes in the breast[s] or nipple[s])

  * History of breast cancer allowed provided ≥ 1 year has elapsed since the last treatment with surgery and there is no known distant metastases and no known residual tumor
* No bilateral breast implants

  * Participants with a unilateral breast implant who would otherwise be eligible for study participation allowed (only breast without implant is evaluated)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 25 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Glomerular filtration rate ≥ 30 mL/min

Other

* Not pregnant or nursing
* Fertile participants must use effective contraception
* Able to undergo adequate mammography and cooperate with breast ultrasound
* No concurrent medical or psychiatric condition that would preclude biopsy
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No contraindications to MRI (e.g., pacemaker, aneurysm clip, or other implanted magnetic device)*
* No claustrophobia that cannot be controlled by medication with valium, ativan, or other sedative*
* Must have intravenous access*
* Weight < 300 pounds*
* Physically able to tolerate positioning in the MRI scanner*
* Able to undergo contrast-enhanced MRI within 4 weeks after completing both study ultrasound and mammogram at 24-month time point*
* Agrees to undergo follow-up MRI at 6 months and/or MRI-guided vacuum-assisted biopsy or ultrasound-guided core biopsy (if needed)* NOTE: *MRI component of the study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy (MRI component of the study)

Endocrine therapy

* See Disease Characteristics
* Concurrent chemoprevention with tamoxifen, raloxifene, anastrozole, exemestane or other aromatase inhibitor for participants with a personal history of cancer allowed (MRI component of the study)

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* More than 1 year since prior fine needle aspiration, core needle biopsy, or surgical procedure
* No prior bilateral mastectomy (MRI component of the study)
* More than 1 year since prior breast surgery on the study breast(s) (MRI component of the study)
* More than 5 months since prior core biopsy of the study breast(s) (MRI component of the study)

Other

* More than 1 year since prior contrast-enhanced MRI of the breast
* More than 1 year (≥ 11 full months) since prior whole breast bilateral ultrasound
* More than 1 year since prior sonographic or mammographic contrast agent injection or tomosynthesis
* More than 2 years since prior screening contrast-enhanced MRI of the study breast(s) (MRI component of the study)
* More than 1 year since prior diagnostic contrast-enhanced MRI of the study breast(s) (MRI component of the study)
* No concurrent participation in any other breast cancer screening trial
* No concurrent participation in any other study involving breast MRI, sonographic or mammographic contrast agents, or tomosynthesis
* No concurrent dialysis

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendie A. Berg, MD, PhD, Study Chair — Johns Hopkins at Green Spring Station
Locations (20):
- United States (18):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Invision - Radiology Imaging Associates, Greenwood Village, Colorado
  - Radiology Associates of Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Johns Hopkins at Green Spring Station, Lutherville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Radiology Consultants, Incorporated, Youngstown, Ohio
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Weinstein Imaging Associates, Pittsburgh, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
- Centro de Estudios Radilogicos Integrales de la Mama - Buenos Aires, Buenos Aires, Argentina
- Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Madsen EL; ACRIN 6666 Investigators. Lesion detection and characterization in a breast US phantom: results of the ACRIN 6666 Investigators. Radiology. 2006 Jun;239(3):693-702. doi: 10.1148/radiol.2393051069. Epub 2006 Apr 26. PMID 16641344
- [Background] Madsen EL, Berg WA, Mendelson EB, Frank GR; Investigators for ACRIN Protocol 6666. Anthropomorphic breast phantoms for qualification of Investigators for ACRIN Protocol 6666. Radiology. 2006 Jun;239(3):869-74. doi: 10.1148/radiol.2393051070. Epub 2006 Apr 26. PMID 16641345
- [Background] Berg WA. Supplemental screening sonography in dense breasts. Radiol Clin North Am. 2004 Sep;42(5):845-51, vi. doi: 10.1016/j.rcl.2004.04.003. PMID 15337420
- [Background] Berg WA. Rationale for a trial of screening breast ultrasound: American College of Radiology Imaging Network (ACRIN) 6666. AJR Am J Roentgenol. 2003 May;180(5):1225-8. doi: 10.2214/ajr.180.5.1801225. No abstract available. PMID 12704027
- [Result] Berg WA, Blume JD, Cormack JB, Mendelson EB. Training the ACRIN 6666 Investigators and effects of feedback on breast ultrasound interpretive performance and agreement in BI-RADS ultrasound feature analysis. AJR Am J Roentgenol. 2012 Jul;199(1):224-35. doi: 10.2214/AJR.11.7324. PMID 22733916
- [Result] Berg WA, Zhang Z, Lehrer D, Jong RA, Pisano ED, Barr RG, Bohm-Velez M, Mahoney MC, Evans WP 3rd, Larsen LH, Morton MJ, Mendelson EB, Farria DM, Cormack JB, Marques HS, Adams A, Yeh NM, Gabrielli G; ACRIN 6666 Investigators. Detection of breast cancer with addition of annual screening ultrasound or a single screening MRI to mammography in women with elevated breast cancer risk. JAMA. 2012 Apr 4;307(13):1394-404. doi: 10.1001/jama.2012.388. PMID 22474203
- [Result] Berg WA, Blume JD, Adams AM, Jong RA, Barr RG, Lehrer DE, Pisano ED, Evans WP 3rd, Mahoney MC, Hovanessian Larsen L, Gabrielli GJ, Mendelson EB. Reasons women at elevated risk of breast cancer refuse breast MR imaging screening: ACRIN 6666. Radiology. 2010 Jan;254(1):79-87. doi: 10.1148/radiol.2541090953. PMID 20032143
- [Result] Berg WA, Sechtin AG, Marques H, Zhang Z. Cystic breast masses and the ACRIN 6666 experience. Radiol Clin North Am. 2010 Sep;48(5):931-87. doi: 10.1016/j.rcl.2010.06.007. PMID 20868895
- [Result] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Derived] Berg WA, Bandos AI, Mendelson EB, Lehrer D, Jong RA, Pisano ED. Ultrasound as the Primary Screening Test for Breast Cancer: Analysis From ACRIN 6666. J Natl Cancer Inst. 2015 Dec 28;108(4):djv367. doi: 10.1093/jnci/djv367. Print 2016 Apr. PMID 26712110